CLINICAL TRIAL: NCT01726400
Title: Is Hepcidin a Possible Contributor to Impaired Iron Mobilization and Anaemia in Hepatitis C Patients Treated With Pegylated Interferon Alpha and Ribavirin Therapy? A Pilot Study
Brief Title: In Hepatitis C Patients Treated With Interferon and Ribavirin, Does Hepcidin Contribute to Treatment Induced Anaemia
Status: Completed | Type: Observational
Sponsor: Fremantle Hospital and Health Service (Other)
Responsible Party: Principal Investigator, Dr Marius van Rijnsoever, Medical Registrar, Fremantle Hospital and Health Service
Other Study IDs: HEPCIDIN-11/225
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Interferon; Ribavirin; Hepcidin; Iron metabolism
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood is collect for genomic DNA extraction. Serum samples will be stored for hepcidin analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Interferon and ribavirin: Treatment with standard of care pegylated interferon alpha and ribavirin.
  Interventions: Drug: Pegylated interferon alpha; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alpha — Subcutaneous weekly pegylated interferon alpha and daily oral ribavirin treatment as per standard treatment. The dosages for interferon and ribavirin are as per therapeutic guidelines and are based on weight, genotype and previous treatments.
  Other Names: pegasys; pegatron
Drug: Ribavirin — Subcutaneous weekly pegylated interferon alpha and daily oral ribavirin treatment as per standard treatment. The dosages for interferon and ribavirin are as per therapeutic guidelines and are based on weight, genotype and previous treatments.
  Other Names: Copegus; Rebetol; Ribasphere; Vilona; Virazole

SUMMARY:
The standard treatment of chronic hepatitis C infection is pegylated interferon alpha combined with ribavirin. Anaemia is a common complication occurring in up to 30% of subjects. Unfortunately, side effects of interferon and ribavirin therapy can require dose reductions, reducing the likelihood of sustained viral response. Recent data shows that interferon alpha may increase hepcidin (a key iron regulator) production, resulting in impaired iron availability for production of red blood cells. In this study, we will evaluate hepcidin levels in 30 patients with Hepatitis C who are treated with interferon containing regimes. If hepcidin plays a role in interferon-induced anaemia, cheap and readily available oral hepcidin inhibitors could be trialled to potentially reduce the impact of interferon alpha induced anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with hepatitis C eligible for treatment with pegylated interferon alpha containing regimes.

Exclusion Criteria:

* less than 18 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C patients undergoing standard of care treatment with interferon alpha.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hepcidin levels | Measured at -2 weeks, start of treatment and week 3,4,8, 12 and 24.
  To measure changes in serum hepcidin levels during pegylated interferon alpha and ribavirin therapy in subjects with chronic hepatitis C infection.

SECONDARY OUTCOMES:
iron metabolism markers | Measured at -2 weeks, start of treatment and week 3,4,8, 12 and 24.
  To measure changes in iron metabolism (reticulocyte haemoglobin, serum iron, transferrin saturation and ferritin levels) during pegylated interferon alpha and ribavirin therapy in subjects with chronic hepatitis C infection.
heamolysis markers | Measured at -2 weeks, start of treatment and week 3,4,8, 12 and 24.
  To detect ribavirin induced heamolysis by measuring serum haptoglobin and free haemoglobin during pegylated interferon alpha and ribavirin therapy in subjects with chronic hepatitis C infection.
inosine triphosphatase genetic variants | Baseline
  To measure the effect of inosine triphosphatase genetic variants on anemia during pegylated interferon alpha and ribavirin therapy in subjects with chronic hepatitis C infection.
erythropoiesis markers | Measured at -2 weeks, start of treatment and week 3,4,8, 12 and 24.
  To measure the level of erythropoiesis (IL1, IL6, erythropoietin and reticulocyte) during pegylated interferon alpha and ribavirin therapy in subjects with chronic hepatitis C infection.

CONTACTS AND LOCATIONS:
Overall Officials: Marius M Van Rijnsoever, MBBS, Principal Investigator — South Metropolitan Health Service, Perth Western Australia
Locations (1):
- Fremantle Hospital, Fremantle, Western Australia, Australia

REFERENCES:
- [Background] Poordad F. Big changes are coming in hepatitis C. Curr Gastroenterol Rep. 2011 Feb;13(1):72-7. doi: 10.1007/s11894-010-0153-9. PMID 21063814
- [Background] Kwo PY, Lawitz EJ, McCone J, Schiff ER, Vierling JM, Pound D, Davis MN, Galati JS, Gordon SC, Ravendhran N, Rossaro L, Anderson FH, Jacobson IM, Rubin R, Koury K, Pedicone LD, Brass CA, Chaudhri E, Albrecht JK; SPRINT-1 investigators. Efficacy of boceprevir, an NS3 protease inhibitor, in combination with peginterferon alfa-2b and ribavirin in treatment-naive patients with genotype 1 hepatitis C infection (SPRINT-1): an open-label, randomised, multicentre phase 2 trial. Lancet. 2010 Aug 28;376(9742):705-16. doi: 10.1016/S0140-6736(10)60934-8. Epub 2010 Aug 6. PMID 20692693
- [Background] Russmann S, Grattagliano I, Portincasa P, Palmieri VO, Palasciano G. Ribavirin-induced anemia: mechanisms, risk factors and related targets for future research. Curr Med Chem. 2006;13(27):3351-7. doi: 10.2174/092986706778773059. PMID 17168855
- [Background] Chua AC, Graham RM, Trinder D, Olynyk JK. The regulation of cellular iron metabolism. Crit Rev Clin Lab Sci. 2007;44(5-6):413-59. doi: 10.1080/10408360701428257. PMID 17943492
- [Background] Olynyk JK, Trinder D, Ramm GA, Britton RS, Bacon BR. Hereditary hemochromatosis in the post-HFE era. Hepatology. 2008 Sep;48(3):991-1001. doi: 10.1002/hep.22507. PMID 18752323
- [Background] Zhang X, Rovin BH. Hepcidin expression by human monocytes in response to adhesion and pro-inflammatory cytokines. Biochim Biophys Acta. 2010 Dec;1800(12):1262-7. doi: 10.1016/j.bbagen.2010.08.005. Epub 2010 Aug 27. PMID 20801192
- [Background] Ward DG, Roberts K, Brookes MJ, Joy H, Martin A, Ismail T, Spychal R, Iqbal T, Tselepis C. Increased hepcidin expression in colorectal carcinogenesis. World J Gastroenterol. 2008 Mar 7;14(9):1339-45. doi: 10.3748/wjg.14.1339. PMID 18322945
- [Background] Ferrari P, Mallon D, Trinder D, Olynyk JK. Pentoxifylline improves haemoglobin and interleukin-6 levels in chronic kidney disease. Nephrology (Carlton). 2010 Apr;15(3):344-9. doi: 10.1111/j.1440-1797.2009.01203.x. PMID 20470305
- [Background] Owen JA, de Gruchy GC, Smith H. SERUM HAPTOGLOBINS IN HAEMOLYTIC STATES. J Clin Pathol. 1960 Nov;13(6):478-82. doi: 10.1136/jcp.13.6.478. PMID 16810960
- [Background] Thompson AJ, Clark PJ, Singh A, Ge D, Fellay J, Zhu M, Zhu Q, Urban TJ, Patel K, Tillmann HL, Naggie S, Afdhal NH, Jacobson IM, Esteban R, Poordad F, Lawitz EJ, McCone J, Shiffman ML, Galler GW, King JW, Kwo PY, Shianna KV, Noviello S, Pedicone LD, Brass CA, Albrecht JK, Sulkowski MS, Goldstein DB, McHutchison JG, Muir AJ. Genome-wide association study of interferon-related cytopenia in chronic hepatitis C patients. J Hepatol. 2012 Feb;56(2):313-9. doi: 10.1016/j.jhep.2011.04.021. Epub 2011 May 20. PMID 21703177
- [Derived] van Rijnsoever M, Galhenage S, Mollison L, Gummer J, Trengove R, Olynyk JK. Dysregulated Erythropoietin, Hepcidin, and Bone Marrow Iron Metabolism Contribute to Interferon-Induced Anemia in Hepatitis C. J Interferon Cytokine Res. 2016 Nov;36(11):630-634. doi: 10.1089/jir.2016.0043. Epub 2016 Sep 12. PMID 27617496
- See also: australian new zealand clinical trials register — http://www.anzctr.org.au/trial_view.aspx?id=347699